CLINICAL TRIAL: NCT02572518
Title: Duration of Immunity After Two Doses of Vaccine Against Yellow Fever in Adults
Brief Title: Immunity After Two Doses of Yellow Fever Vaccine
Acronym: IATDYFV
Status: Completed | Type: Observational
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Responsible Party: Sponsor
Other Study IDs: ASCLIN 003/2013
Record Dates: First submitted 2015-09-16; First posted 2015-10-09 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Yellow Fever
Keywords: immunity yellow fever vaccine
MeSH Terms: conditions — Yellow Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 45 Days
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 2 doses of yellow fever vaccine: 30 days,1-5 years and 6 years or more after last dose

SUMMARY:
To evaluate the immune status of yellow fever in adults with a history of two or more doses of vaccine, having received the second dose for at least 1 year, compared to re-vaccinated individuals (second dose) after 30 days.

DETAILED DESCRIPTION:
Data Collection Volunteers will be invited to participate by bringing card (s ) vaccination or copy ( s ) of record ( s ) in which it appears ( m) ( s ) dose ( s) received yellow fever vaccine ( s ) and ( s ) their ( s ) date ( s ) . Individuals who agree to participate in the study and signed an Informed Consent Form will be forwarded to interview and application of Inclusion Questionnaire , which will identify possible eligible for the study and classify them according to the time of vaccination. Then a medical review of the history of vaccination with the date or the age in which they occurred , the cities and the period in which he lived and the relevant pathological history , hospitalizations and treatment for chronic diseases will be taken , then proceeding to blood collection.

Upon completion of the subject's participation in the research study , registration must be done at the closing to participate in the study .A group of volunteers previously vaccinated with a dose of yellow fever vaccine and booster having the indicated activity in the areas in which the vaccine is recommended that , constitute a group of 110 patients with different to the search approach, in which a pickup is performed Whole blood for analysis of cellular immune 30-45 days after revaccination.

The clinical forms of the study will be prepared and processed in " TELEform " program , which will enable the digitization and preparation of database.

Sample Size Whereas 98% seropositivity and presence of cellular response after 30 days of revaccination as reference, 110 volunteers will be needed in each group to detect minute differences of 10 percentage points with 80% power and a significance level of 5%.

A total of 440 volunteers with 110 distributed in each group. Samples of 110 individuals will estimate proportions of seropositive up to 50% with precision of 9 percentage points for each side.

Biological Samples Samples are initially obtained from 10 ml of peripheral blood collected without anti-coagulant for serology, in all volunteers (N = 440).

For a subset of 200 subjects (50 in each group) are also collected 20 ml of blood in heparin (10 mL of 2 tubes) for determination of cellular immunity. Specifically for the reference group, the collection of 20ml will be held at two different times, the first visit and return visit, 30 to 45 days after revaccination.

Laboratory tests Titration of neutralizing antibodies ( PRNT ):the neutralizing antibody titers of volunteers will be determined by neutralization test for 50% reduction of plaques of lysis buffer ( PRNT50 ) in monolayers of Vero cells.

For neutralization tests PRNT by the dosage of antibody is expressed in milli- International Units per milliliter ( mlU / ml) of serum.

In a subsample of 20 % of individuals, subalíquota serum will be separated to be reviewed with the PRNT for yellow fever in order to allow verification that the serological tests performed by another team .

ELISA:Serological tests ( IgG ) for dengue will be held . These same samples will be tested for IgG -ELISA for confirmation of antiamarílicos antibodies in the sera of vaccinated people. Additionally , the level of IgG antibodies in the serum by a conventional method collected from volunteers to compare the data from literature is performed.

Presence of cellular immunity: Aliquots of 20 mL of whole blood is collected into tubes containing sodium heparin anticoagulant ( Vacutainer , BD , USA ) for the culture of peripheral blood mononuclear cells (PBMC ).

Monitoring of adverse events As the administration of vaccines is not a research activity, the record of the post-vaccination adverse events should be done by professionals who administer the vaccine in accordance with the Manual of Epidemiological Surveillance of Adverse Events Following Immunization, 2nd. Edition - 2009, Ministry of Health, research and monitoring of post-yellow fever vaccination serious adverse events, the Ministry of Health

Statistical Analysis The response variable of interest is the titer of neutralizing antibodies ( in mIU / mL ) of serum and transformed into logarithms base 10 . The serological status variable will be derived - seropositive : antibody titers of equal to or greater than 2.8 log10 mIU / mL ; seronegative : securities equal to or less than 2.6 log10 mIU / mL, and indeterminate : securities equal to 2.7 log10 mIU / mL .

The proportion of seropositivity and geometric mean antibody titers are estimated ( with their corresponding 95 % confidence ) for each study group : revaccinated for 30 days vaccinated with two doses there 1-5 years, 6 years or more vaccinated with three doses or more .

The seropositivity and the profile of cellular immunity in the subgroup of individuals revaccinated thirty days will be taken as reference for comparisons with other groups . The serological and cellular immunity in this subgroup profile before the second vaccination will also be used as a reference for comparisons.

The covariates for analysis are: age (continuous variable in years) the last dose of yellow fever vaccine, sex, presence of antibodies against dengue vaccination history, history of severe illness (hospitalization, sequelae, disability) and co-morbidity (who used drugs at the time of blood sampling).

ELIGIBILITY:
Inclusion Criteria:

-Will be eligible for the study volunteers with proof of vaccination in vaccine design or functional or health care records, and who agree to participate in the study.

Exclusion Criteria:

-Will not be included adults with a contraindication for vaccination against Yellow Fever (permanent or transient immunosuppression, severe adverse reaction after the first dose, severe allergy to chicken eggs), use of hyperimmune serum or vaccine within 30 days prior to collection blood, individuals without proof (s) of vaccination (s) above (ies) or individuals who have resided or traveled to endemic or considered risk areas by the Ministry of Health, regardless of length of stay in high-risk areas.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The target study population will consist of 440 adult who have previously received at least one dose of yellow fever 17DD vaccine. The volunteers who received two doses of vaccine will be distributed in subgroups 1-5 and 6 years old or more, relative to the date of the last dose received. Volunteers with just one dose and who have received the same for at least 10 years, constitute the reference group (control) for serological and immunological studies. These volunteers will be guided and directed to revaccination in rooms vaccine immunization program and 30 to 45 days after revaccination shall be subjected to serological testing.
Sampling Method: Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Access the change of the immune status to yellow fever in adults history of two or more doses of vaccine, having received the second dose for at least one year, compared to revaccinated individuals (second dose) after 30 days. | 30 days, 1-5 years, through study completion at least 6 years after second dose of yellow fever vaccine, with 3 doses at any age

SECONDARY OUTCOMES:
Access the cellular immunity | 30 days, 1-5 years, through study completion at least 6 years after second dose of yellow fever vaccine, with 3 doses at any age
  Evaluating and comparing through inmunofenotípica characterization of markers cell surface, the frequency of T lymphocytes (CD4, CD27, CD8, CD45RO, CD183 (CXCR3), CD3) and B (CD27, CD19, CD38, CD10, CD3) memory, in vitro induced by the vaccine antigen 17DD in adults with at least two doses of vaccine in each group

OTHER OUTCOMES:
Access the cellular immunity | 30 days, 1-5 years,through study completion at least 6 years after second yellow fever vaccine, with 3 doses at any age
  Dosing and comparing by flow cytometry, intracytoplasmic cytokines (CD8 + subpopulations of T lymphocytes, IFN-gamma, IL-5, TNF-alpha) and soluble (IFNalpha, IFN-gamma, TNF-alpha, IL-4, IL-5 and IL-10) in adults with two or more vaccine doses, categorized according to the time since the last dose: 30 days 1-5 years, 6 years or more
Access the cross reaction humoral immune status (neutralizing antibody) and cellular (aspects functional and phenotypic) | 30 days, 1-5 years,through study completion at least 6 years after second yellow fever vaccine, with 3 doses at any age
  Evaluating the influence of exposure to dengue virus IgG antibodies anti-in humoral immune status (neutralizing antibody) and cellular (aspects functional and phenotypic) in adults with two or more doses of vaccine, categorized according to the time since the last dose: 30 days, 1-5 years, through study completion at least 6 years and with 3 doses.

CONTACTS AND LOCATIONS:
Overall Officials: T G N, Principal Investigator — Institute of Technology in Immunobiology Bio-Manguinhos/Fiocruz
Locations (1):
- Institute of Technology in Immunobiology Bio-Manguinhos/Fiocruz, Rio de Janeiro, Rio de Janeiro, Brazil